CLINICAL TRIAL: NCT04066205
Title: Sleep Shared-Management Intervention for Children With Juvenile Idiopathic Arthritis
Acronym: SLEEPSMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Teresa Ward, Professor, School of Nursing: Psychosocial and Community Health, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00005070; R21NR017471-01A1 (NIH)
Record Dates: First submitted 2018-09-05; First posted 2019-08-26 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-12

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Sleep deficiency, self-management
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Intervention Model Description: This pilot RCT, comparing usual care to SLEEPSMART intervention with 60 JIA children and their parents
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SLEEPSMART PROGRAM (Experimental): Arm: Placebo Comparator (Usual care)-This treatment arm will receive usual JIA care, including annual Rheumatology clinic visits, medications, routine clinical and laboratory tests, physical therapy, follow-up appointments, and no sleep intervention.
  Arm: Experimental -Each child and parent dyad will work together to create sleep goals, problem solve and compromise to accomplish the goals, and interact with fields in the Web site. The modules will focus on learning a wind-down and wake-up routine, reducing time in bed, reducing sleep-related worry, negotiating sleep in the environment, correcting unhelpful sleep-related beliefs, and sleep maintenance and relapse prevention. The intervention will last 7 weeks.
  Interventions: Behavioral: SLEEPSAMRT

INTERVENTIONS:
Behavioral: SLEEPSAMRT — SLEEPSMART is a web-based intervention that adapted and modified components from the Transdiagnostic Sleep and Circadian intervention for youth and included four cross-cutting components (sleep complaint, education, behavior change and motivation, and goal-setting) that were integrated into each module. To begin the intervention, participants were provided a link to the SLEEPSMART intervention website for one of the above modules and an online sleep coach each week. At the end of each week, children and parents uploaded the weekly activities and goals via the REDCap link and set up a meeting with the sleep coach to review. The modules took 20 to 30 minutes to complete.

SUMMARY:
Sleep deficiency is a public health concern in children with a chronic illness such as Juvenile Idiopathic Arthritis (JIA) because it is often overlooked in clinical care, attributed to the underlying chronic illness, and contributes to poor health outcomes. Development of an effective technology-based sleep shared-management intervention that integrate children and parents in the co-design and development of the intervention has the potential to improve health outcomes of children living with JIA and their parents.

DETAILED DESCRIPTION:
To develop and test a technology-based sleep shared-management intervention delivered to 8-to-13 year-old children with JIA and their parents. The initial feasibility, acceptability, and efficacy of the newly developed sleep shared-management intervention will be tested in a pilot randomized controlled trial comparing the active intervention against standard care with a sample of 60 children with JIA and their parents. Sleep will be measured using actigraphy, sleep diaries, & self-report measures. Self-efficacy will be measured before and after the intervention. The long-term goal is to develop effective and low cost treatments to reduce sleep deficiency and the sleep-related health consequences among children with JIA. The specific aims are to:

Aim 1. Apply a human-centered design approach to develop and refine a technology-based sleep shared-management intervention (SLEEPSMART). Direct stakeholder input will be obtained from children and parents about their needs for sleep shared-management as well as intervention material adapted from the Transdiagnostic Sleep-Circadian Dysfunction program for youth that includes four cross cutting components (sleep complaint, education, behavior change and motivation, and goal setting) across the modules and a shared- management focus (motivation, self-efficacy) with children and parent partnering together to improve sleep. Qualitative methods (iterative cycles of semi-structured audiotaped sessions with children and parents and think-aloud observation sessions by a trained observer) will be used to evaluate the usability of the SLEEPSMART prototype. Results of these analyses will guide program finalization.

Aim 2. Determine feasibility and initial efficacy of the SLEEPSMART with children with JIA in a pilot RCT. Study accrual and dropout rates will be assessed, as well as, levels of patient acceptability and engagement in a pilot randomized controlled trial (RCT) comparing usual care to SLEEPSMART intervention. Preliminary effect sizes of the SLEEPSMART will be determined in youth receiving treatment compared to usual care on primary outcomes of actigraphy sleep duration, self-report sleep disturbances, and feasibility/acceptability, and secondary outcomes include self-efficacy.

ELIGIBILITY:
Inclusion Criteria for Children:

* diagnosed with JIA, 8-13 years, and parent report that child has difficulties with sleep quality (difficulty falling asleep, no bedtime routine, waking up in the middle of the night and struggling to fall back asleep) and/or poor sleep impacts their child's day to day function (school, interacting with peers, hobbies).

Inclusion criteria for parents:

* > 18 years, access to a computer or web-based device to complete the surveys, and residing with the child more than 50% of the time

Exclusion Criteria for Children:

* Diagnosed with a sleep disorder (OSA), positive screen on the pediatric sleep questionnaire for OSA, lack of daily access to the internet, developmental delay, currently taking sleep medication (melatonin), and currently participating in psychological therapy and/or participated in psychological therapy the prior 3 months.

Exclusion criteria for parents:

* diagnosed with a chronic illness that would interfere with ability to complete study procedures

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa M Ward, RN, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington School of Nursing, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhai S, Palermo TM, Shenoi S, Demiris G, Howard W, Kientz J, Yuwen W, Ward TM. A shared-management web-based intervention for sleep deficiency in school-age children with juvenile idiopathic arthritis and their parents: feasibility and acceptability study. J Clin Sleep Med. 2025 Jun 1;21(6):1007-1021. doi: 10.5664/jcsm.11610. PMID 40051205

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 50 children with JIA and 50 parents.
Pre-assignment Details: The number of participants in each Milestone represents each child and each parent in the SLEEPSMART Intervention group and each child and each parent in the control group.
Groups:
- SLEEPSMART PROGRAM: Arm: Experimental -Each child and co-parent dyad will work together to create sleep goals, problem solve and compromise to accomplish the goals, and interact with fields in the Web site. The weekly modules will focus on learning a wind-down and wake-up routine, reducing time in bed, reducing sleep-related worry, negotiating sleep in the environment, correcting unhelpful sleep-related beliefs, and sleep maintenance and relapse prevention. The intervention will last 7 weeks.
- Placebo Comparator (Usual Care): Arm: Placebo Comparator (Usual care)-This treatment arm will receive usual JIA care, including annual Rheumatology clinic visits, medications, routine clinical and laboratory tests, physical therapy, follow-up appointments, and no sleep intervention.
Period: Baseline
Arm/Group | SLEEPSMART PROGRAM | Placebo Comparator (Usual Care)
Started | 50 (50 represents each child and each parent.) | 50 (50 represents each child and each parent.)
Completed | 48 (48 represents EACH child and EACH parent) | 40 (40 represents each child and each parent.)
Not Completed | 2 | 10
Period: T2 Immediate Post-Intervention
Arm/Group | SLEEPSMART PROGRAM | Placebo Comparator (Usual Care)
Started | 48 (48 represents each child and each parent) | 40 (40 represents each child and each parent.)
Completed | 38 (38 represents each child and each parent.) | 34 (34 represents each child and each parent dyad.)
Not Completed | 10 | 6
Not completed — Did not respond during intervention or usual care | 5 | 3
Not completed — did not respond | 5 | 3
Period: T3 One Month Post-Intervention
Arm/Group | SLEEPSMART PROGRAM | Placebo Comparator (Usual Care)
Started | 38 (38 represents each child and each parent.) | 34 (34 represents each child and each parent)
Completed | 38 (38 represents each child and each parent.) | 34 (34 represents each child and each parent)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants reflect EACH child and parent( for the SLEEPSMART program 24 dyads child /co-parent dyads received the SLEEPSMART intervention; and 20 children with JIA and their co-parent were in the control group.
Groups:
- SLEEPSMART PROGRAM: Arm: Experimental group 24 children and 24 parents (n=48) that equates to 24 child/co-parent dyads
- Placebo Comparator (Usual Care): Arm: Placebo Comparator (Usual care) represents 20 children and 20 parents (n=40) that equates to 20 child/co-parent dyads. This treatment arm will receive usual JIA care, including annual Rheumatology clinic visits, medications, routine clinical and laboratory tests, physical therapy, follow-up appointments, and no sleep intervention.
- Total: Total of all reporting groups
Arm/Group | SLEEPSMART PROGRAM | Placebo Comparator (Usual Care) | Total
Number analyzed (Participants) | 48 | 40 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] — Child age Population: This represent EACH child and EACH parent in SLEEPSMART Group AND Control Group.
  years
    Child: number analyzed (Participants) | 24 | 20 | 44
    Child | 10.1 (1.7) | 10.5 (1.8) | 10.3 (1.7)
    Parent: number analyzed (Participants) | 24 | 20 | 44
    Parent | 40.7 (5.4) | 43.3 (6) | 41.95 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants] — Child gender Population: These numbers represent EACH child and parent
  Participants
    Child: number analyzed (Participants) | 24 | 20 | 44
    Child: Female | 18 | 18 | 36
    Child: Male | 6 | 2 | 8
    Parent: number analyzed (Participants) | 24 | 20 | 44
    Parent: Female | 24 | 20 | 44
    Parent: Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Child Ethnicity Population: These numbers represent EACH child and parent
  Participants
    Child: number analyzed (Participants) | 24 | 20 | 44
    Child: Hispanic or Latino | 4 | 6 | 10
    Child: Not Hispanic or Latino | 20 | 14 | 34
    Child: Unknown or Not Reported | 0 | 0 | 0
    Parent: number analyzed (Participants) | 24 | 20 | 44
    Parent: Hispanic or Latino | 4 | 5 | 9
    Parent: Not Hispanic or Latino | 20 | 15 | 35
    Parent: Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Child race Population: These numbers represent EACH child and parent.
  Participants
    Child: number analyzed (Participants) | 24 | 20 | 44
    Child: American Indian or Alaska Native | 0 | 0 | 0
    Child: Asian | 0 | 0 | 0
    Child: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Child: Black or African American | 0 | 0 | 0
    Child: White | 20 | 17 | 37
    Child: More than one race | 2 | 2 | 4
    Child: Unknown or Not Reported | 2 | 1 | 3
    Parent: number analyzed (Participants) | 24 | 20 | 44
    Parent: American Indian or Alaska Native | 0 | 0 | 0
    Parent: Asian | 0 | 0 | 0
    Parent: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Parent: Black or African American | 0 | 0 | 0
    Parent: White | 21 | 17 | 38
    Parent: More than one race | 3 | 3 | 6
    Parent: Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Sleep Disturbance
Description: PROMIS Sleep Disturbance an 8-item questionnaire that measures self-reported perceptions of sleep quality, depth, and restoration within the past seven days. Items are rated on a 5-point Likert scale (1= not at all/very poor, 2 = a little bit/poor, 3=somewhat/fair, 4=quite a bit/good, 5= very much/very good). The raw scores are converted into a T-score. The T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Higher T-scores suggest more disturbed sleep.
Time Frame: Baseline (start of the study); 2 months (immediately after the intervention), and 3 months (study completion)
Population: At 2 and 3 months, some participants could not be reached or declined to participate.
Measure: Mean (Standard Deviation); unit: T-score
Groups:
- SLEEPSMART PROGRAM: Arm: Experimental -Each child and parent will partner with a sleep coach each week to review their weekly goals and choose new treatment goals. The modules will focus on improving wind down and wake up routine, sleep hygiene, relaxation techniques, correcting unhelpful sleep beliefs, and changing the sleep environment. The intervention will last 7 weeks.
Arm/Group | SLEEPSMART PROGRAM | Placebo Comparator (Usual Care)
Number analyzed (Participants) | 24 | 20
T-score
  Baseline | 62.1 (5.4) | 62.4 (7.3)
  2 months: number analyzed (Participants) | 19 | 17
  2 months | 57.7 (4.3) | 58.3 (7.6)
  3 months: number analyzed (Participants) | 19 | 17
  3 months | 56.4 (2.8) | 58.5 (7.1)

2. Primary Outcome: Sleep Efficiency
Description: Actigraphy variable defined as the ratio of total sleep time/time in bed where 1.0 is the most efficient sleep.
Time Frame: Baseline (start of the study); 2 months (immediately after the intervention), and 3 months (study completion)
Population: At 2 months and 3 months, some participants declined to participate or could not be reached.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | SLEEPSMART PROGRAM | Placebo Comparator (Usual Care)
Number analyzed (Participants) | 24 | 20
ratio
  Baseline | .74 (.08) | .78 (.05)
  2 months: number analyzed (Participants) | 19 | 17
  2 months | .83 (.05) | .79 (.04)
  3 months: number analyzed (Participants) | 19 | 17
  3 months | .84 (.07) | .79 (.04)

3. Primary Outcome: Sleep Duration
Description: Actigraphy variable Total Sleep Time (TST), defined as the minutes during the sleep period;
Time Frame: baseline (start of the study); 2 months (immediately after the intervention) and 3 months (study completion)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | SLEEPSMART PROGRAM | Placebo Comparator (Usual Care)
Number analyzed (Participants) | 24 | 20
minutes
  Baseline | 464.0 (46.7) | 483.2 (25.1)
  2 months | 508.6 (57.4) | 483.6 (28.1)
  3 months | 506.7 (48.1) | 488.7 (33.4)

4. Primary Outcome: Acceptability of SLEEPSMART
Description: Parent and child survey about the likes and dislikes of the study protocol, areas for improvement, SLEEPSMART program and weekly assignments. Items are scored using a 5-point scale, with 1 equalling strongly disagree and 5 equalling strongly agree. Scores can range from 9 to 45 with higher scores representing greater acceptance. A total score of moderate acceptability for the nine items would be 27.
Time Frame: 3 months at study completion
Population: At 2 months and 3 months, some participants declined to participate or could not be reached.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SLEEPSMART Child; SLEEPSMART Parent: SLEEPSMART will be designed to improve sleep by providing guidance and structure to assist JIA children and their parent in adhering to the intervention protocol. The intervention will be interactive and personalized; users will interface with three primary components:1) monitoring: daily records of sleep and symptoms; 2) skill building modules: sleep education, sleep skills training, relaxation techniques, positive coping skills, and reward systems for activity participation for reducing sleep deficiency; and 3) assignment review and personalized feedback via behavioral assignments for skill implementation and tailored feedback. Modules will take an estimated 30 minutes each week to complete and will include multimedia elements to enhance learning.
Arm/Group | SLEEPSMART Child | SLEEPSMART Parent
Number analyzed (Participants) | 12 | 12
score on a scale | 34.1 (8.2) | 36.6 (6.4)

5. Secondary Outcome: Self-efficacy Child
Description: Self-Efficacy scale: 9-item self-report of confidence in carrying out sleep-related behaviors; Likert scale from 1 (not at all confident) to 10 (totally confident); higher score indicates better self-efficacy.
Time Frame: Baseline (start of the study); 2 months (immediately after the intervention) and 3 months (study completion)
Population: At 2 months and 3 months, subjects (3 Placebo and 5 SLEEPSMART Intervention) declined to participate or could not be reached.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- SLEEPSMART PROGRAM: Arm: Experimental -Each child and parent will create a login, choose treatment goals, and interact with fields in the Web site. The modules will focus on improving sleep hygiene, relaxation, or increasing sleep duration. The intervention will last 6 to 8 weeks.
Arm/Group | SLEEPSMART PROGRAM | Placebo Comparator (Usual Care)
Number analyzed (Participants) | 24 | 20
score on a scale
  Baseline | 2.5 (.8) | 2.4 (2.8)
  2 Months: number analyzed (Participants) | 19 | 17
  2 Months | 2.0 (.6) | 2.3 (.8)
  3 Months: number analyzed (Participants) | 19 | 17
  3 Months | 2.0 (.8) | 2.2 (.9)

6. Secondary Outcome: Self-efficacy Parent
Description: A 9-item survey that assesses parent confidence to manage/control their children's chronic conditions and sleep, emotional functioning, and communication with healthcare providers. Items are rated using a visual analog scale, ranging from 1 = not at all confident to 10 = totally confident. A mean score is calculated with higher values indicative of higher self-efficacy
Time Frame: baseline (start of the study); 2 months (immediately after the intervention) and 3 months (study completion)
Population: At 2 months and 3 months, some particpants declined to participate or could not be reached.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SLEEPSMART PROGRAM | Placebo Comparator (Usual Care)
Number analyzed (Participants) | 24 | 20
score on a scale
  Baseline | 5.8 (1.9) | 6.5 (1.6)
  2 months: number analyzed (Participants) | 19 | 17
  2 months | 7.1 (1.3) | 6.6 (1.9)
  3 months: number analyzed (Participants) | 19 | 17
  3 months | 7.5 (1.4) | 7.2 (1.9)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 3 months.
Description: Parents/caregiver and children adverse events reporting were combined by dyad since parents and children were enrolled by dyad. It was a shared management intervention where parents partnered with children and the majority of data was obtained via surveys that are typically low risk for adverse events.
Groups:
- SLEEPSMART PROGRAM: Arm: Experimental -Each child and parent will partner with a sleep coach to review weekly goals and choose treatment goals. The modules will focus on improving wind down and wake up routines, sleep hygiene, relaxation strategies, correcting unhelpful beliefs about sleep, and the sleep environment. The intervention will last 7 weeks..
Arm/Group | SLEEPSMART PROGRAM | Placebo Comparator (Usual Care)
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/21
Other Adverse Events (participants affected / at risk) | 0/25 | 0/21

LIMITATIONS AND CAVEATS:
1. Single-site pilot trial which may limit the generalizability of the findings.
2. Our follow-up period was limited to one-month post-intervention, and some children and parents may have needed a longer time to see the effects of SLEEPSMART.
3. Study was conducted during the COVID-19 pandemic, and stay-at-home guidance may have altered sleep routines and patterns for children and parents.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-23): https://cdn.clinicaltrials.gov/large-docs/05/NCT04066205/Prot_SAP_000.pdf